CLINICAL TRIAL: NCT04299438
Title: Propranolol Rescue of Prolonged Labor (PROPEL): A Randomized, Double-blind, Placebo-controlled Multicenter Investigation of Propranolol's Effect on Cesarean Delivery Rate Among Women With Prolonged Labor
Brief Title: Propranolol Rescue of Prolonged Labor
Acronym: PROPEL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped at interim analysis
Sponsor: Lisa Levine (Other)
Responsible Party: Sponsor-Investigator, Lisa Levine, Assistant Professor of Obstetrics and Gynecology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 834760
Record Dates: First submitted 2020-02-25; First posted 2020-03-06 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy, Prolonged
Keywords: Propranolol; Cesarean
MeSH Terms: conditions — Pregnancy, Prolonged | interventions — Propranolol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propranolol (Active Comparator): IV Propranolol - 2mg; one possible repeat dose ≥2 hours later
  Interventions: Drug: Propranolol Hydrochloride
- Placebo (Placebo Comparator): Normal saline placebo- 2 mL; one possible repeat dose ≥2 hours later
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Propranolol Hydrochloride — 2mg/mL vials
  Other Names: Inderal
  Arms: Propranolol
Other: Saline — 0.9% saline in vials matching the vials of the active drug
  Arms: Placebo

SUMMARY:
A double-blind placebo controlled randomized trial comparing cesarean delivery rates in women given IV propranolol versus placebo for treatment of prolonged labor.

DETAILED DESCRIPTION:
A double-blind placebo controlled randomized trial comparing cesarean delivery rates in 326 women given IV propranolol (2 mg with one possible repeat dose greater than 2 hours later) versus IV placebo for treatment of prolonged labor.

ELIGIBILITY:
Inclusion Criteria:

English-speaking

>= 36 weeks gestation

Singleton pregnancy

Vertex presentation

No contraindication to a vaginal delivery

Meets at least one study criteria for prolonged labor:

1. cervical dilation <6 cm after ≥8 hours with ruptured membranes and receiving oxytocin OR
2. cervical dilation >=6 cm and <1 cm dilation change over ≥2 hours with ruptured membranes and receiving oxytocin

Exclusion Criteria:

Severe preeclampsia: as patients will be receiving magnesium and possibly labetalol for hypertension control

Receiving other beta blocker

Maternal heart rate < 70 beats per minute, systolic blood pressure <90 mmHg, or diastolic blood pressure <50 mmHg on two sets of vital signs in the 1 hour prior to study drug administration: given that bradycardia and hypotension are possible side effects of propranolol

History of any form of asthma: as this is a contraindication to beta blocker use

Diabetes requiring insulin in labor: given the potential risk of neonatal hypoglycemia in the neonate

Any cardiac condition for which β blockade is contraindicated (cardiogenic shock, sinus bradycardia, and greater than first degree heart block)

Known hypersensitivity to propranolol

Intrauterine fetal demise since different labor protocols are used in these women

Major fetal congenital anomaly since rate of cesarean may be inherently different in these women, unrelated to labor

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Levine, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCoy JA, Walheim L, McCabe MG, Levine LD. Efficacy of Propranolol to Reduce Cesarean Delivery in Prolonged Labor: A Randomized Controlled Trial. Obstet Gynecol. 2023 Jul 1;142(1):71-79. doi: 10.1097/AOG.0000000000005232. Epub 2023 Jun 7. PMID 37290102

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Post-enrollment exclusion: if patient made cervical change or delivered after enrollment but prior to randomization
Period: Overall Study
Arm/Group | Propranolol | Placebo
Started | 84 | 80
Completed | 84 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: trial stopped by DSMB after interim analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Placebo | Total
Number analyzed (Participants) | 84 | 80 | 164
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29.3 [23.4 to 32.6] | 30.1 [22.8 to 33.2] | 29.4 [23.1 to 32.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 80 | 164
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 49 | 98
  White | 33 | 23 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 8 | 10
Region of Enrollment [Number; unit: participants]
  United States | 84 | 80 | 164

OUTCOME MEASURES:

1. Primary Outcome: Mode of Delivery
Description: Number of participants with a cesarean delivery
Time Frame: From enrollment into the trial until delivery.
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 84 | 80
Participants | 48 | 46

2. Secondary Outcome: Length of Labor
Description: Time in hours from start of labor or induction of labor to delivery
Time Frame: hours from start of labor or induction of labor to time of delivery
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 84 | 80
hours | 26.6 [20.6 to 34.3] | 28.4 [24.1 to 32.2]

3. Secondary Outcome: Postpartum Hemorrhage
Description: Amount of blood loss measured in mL
Time Frame: from time of delivery through hospital discharge, usually 2-4 days
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 84 | 80
Participants | 17 | 8

4. Secondary Outcome: Chorioamnionitis
Description: Number of participants with chorioamnionitis
Time Frame: from start of labor through delivery
Population: intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 84 | 80
Participants | 18 | 24

5. Secondary Outcome: Maternal Morbidity
Description: Number of participants with 1 or more of the following: blood transfusion, endometritis, wound infection, venous thromboembolism, hysterectomy, ICU admission, readmission, death
Time Frame: from delivery through 4 weeks postpartum
Population: intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 84 | 80
Participants | 10 | 5

6. Secondary Outcome: Neonatal Morbidity
Description: Number of participants with 1 or more of the following: Intensive care nursery admission >48, blood transfusion, hypoxic-ischemic encephalopathy, intraventricular hemorrhage grade 3 or 4, neonatal head cooling, severe respiratory distress syndrome, necrotizing enterocolitis, sepsis, death
Time Frame: from delivery through hospital discharge, usually 2-4 days
Population: intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 84 | 80
Participants | 7 | 4

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Propranolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/80
Serious Adverse Events (participants affected / at risk) | 3/84 | 1/80
Other Adverse Events (participants affected / at risk) | 46/84 | 46/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=84) | Placebo (N=80)
Neonataly hypoxic ischemic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Intensive care unit admission (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Maternal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Anaphylaxis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Hysterectomy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Neonatal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Neonatal blood transfusion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Neonatal intraventricular hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Neonatal severe respiratory distress (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Necrotising enterocolitis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Culture proven neonatal sepsis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=84) | Placebo (N=80)
Neonatal hypoglycemia (Endocrine disorders) | 24 (24) | 20 (20)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 18 (18) | 24 (24)
Endometritis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Venous thromboembolism (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Readmission within 7 days (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
NICU admission >48 hours (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 4 (4)
Maternal bradycardia <50 beats per minute within 30 minutes of drug administration (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Maternal hypotension <80/40 mmHg within 30 minutes of drug administration (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Maternal bronchospasm (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Maternal hypoglycemia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)
Allergic reaction (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT04299438/Prot_SAP_003.pdf